CLINICAL TRIAL: NCT02525497
Title: A Randomized, Multicenter, Crossover Study Comparing the Domestic FM Peritoneal Dialysis Machine With Baxter HOMECHOICE
Brief Title: Safety, Effectiveness and Manipulability Evaluation of a Domestic PD Machine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiangmei, professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MD-PD-2014
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Kidney Failure,Chronic
Keywords: Automated PD; Effectiveness; Safety; Manipulability
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FM peritoneal dialysis machine (Experimental): FM peritoneal dialysis machine APD 10L/10h;
  Interventions: Device: FM peritoneal dialysis machine
- HOMECHOICE peritoneal dialysis machine (Active Comparator): HOMECHOICE peritoneal dialysis machine APD 10L/10h;
  Interventions: Device: HOMECHOICE peritoneal dialysis machine

INTERVENTIONS:
Device: FM peritoneal dialysis machine — FM peritoneal dialysis machine APD 10L/10h
  Arms: FM peritoneal dialysis machine
Device: HOMECHOICE peritoneal dialysis machine — HOMECHOICE peritoneal dialysis machine APD 10L/10h
  Arms: HOMECHOICE peritoneal dialysis machine

SUMMARY:
This study is a randomized, multi-center，crossover study of a domestic FM peritoneal dialysis machine and Baxter HOMECHOICE.It aims to verify safety, effectiveness and manipulability of a domestic peritoneal dialysis machine.

DETAILED DESCRIPTION:
Our study is a randomized, multi-center，crossover study. It compares a domestic FM peritoneal dialysis machine with Baxter HOMECHOICE.It aims to verify safety, effectiveness and manipulability of a domestic peritoneal dialysis machine.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18, male or female Dialysis duration:≥30 days Sign the written informed consent

Exclusion Criteria:

Hemodialysis Exit site infection or tunnel infection Peritonitis ≤30 days before screening Catheter mechanical failure Anti-HIV positive Allergic to components of dialysate Comorbidity:Active, residual malignant tumor, or systemic infection, liver cirrhosis, severe congestive heart failure,hypertension Poor compliance Pregnant or lactating, women of childbearing age do not agree to use effective contraceptive measures during the trial Has a history of alcoholism and drug abuse (defined as illegal drugs) Any circumstances when patients are believed unsuitable for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Daily peritoneal Kt/V | 1 day

SECONDARY OUTCOMES:
The accuracy of filling | 1 day

OTHER OUTCOMES:
The accuracy of filling temperature | 1 day
Serum sodium before and after dialysis | 1 day
Serum potassium before and after dialysis | 1 day
Serum calcium before and after dialysis | 1 day
Serum phosphorus before and after dialysis | 1 day
Serum carbon dioxide binding force before and after dialysis | 1 day
Serum creatinine before and after dialysis | 1 day
Serum urea nitrogen before and after dialysis | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: CHEN Xiangmei, yes, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao XY, He YN, Zhou JH, Sun SR, Miao LN, Chen W, Fang JA, Wang M, Wang NS, Lin HL, Liu J, Ni ZH, Liu WH, Na Y, Zhao JY, Guo ZY, Zheng HG, Shi W, Jiang GR, Cai GY, Chen XM. Safety, Effectiveness, and Manipulability of Peritoneal Dialysis Machines Made in China: A Randomized, Crossover, Multicenter Clinical Study. Chin Med J (Engl). 2018 Dec 5;131(23):2785-2791. doi: 10.4103/0366-6999.246079. PMID 30511680